CLINICAL TRIAL: NCT05896878
Title: The Effects of Daily Anti-inflammatory Supplementation on Foundation Pain Index Scores in Chronic Opiate Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Product terminated
Sponsor: Hudson Medical (Other)
Collaborators: Ethos Research & Development (Industry)
Responsible Party: Principal Investigator, Jonathann Kuo, MD, Principial Investigator, Hudson Medical
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRANY #22-02-797-993
Record Dates: First submitted 2023-04-07; First posted 2023-06-09 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Pain, Chronic; Opioid Dependence; Opioid Use; Inflammation Chronic
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: This study is a prospective, open-label, non randomized evaluation of daily supplementation with Root.Health, a plant-based anti-inflammatory dietary supplement, on Foundation Pain Index (FPI) scores in a chronic opiate patient population. The daily supplement is offered without charge to study participants. All patients are counseled and consented per established protocol as per established IRB requirements. This study will enroll 20 total patients. The details of the study design, patient demographics, description of the intervention method, and statistical tests performed are described.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Daily Supplement Treatment (Experimental): Following study recruitment and obtaining consent, participants will complete a baseline urine test. The FPI is a simple urine test from Ethos Laboratories that screens for 11 biomarkers that are more likely to contribute to symptoms of pain.
  Interventions: Dietary Supplement: Root.Health Dietary Supplement

INTERVENTIONS:
Dietary Supplement: Root.Health Dietary Supplement — The Root.Health supplement is composed of six plant-based compounds with established roles in supporting innate physiological processes which are implicated in pain: tetrohydrocurcumin, ergothioneine, dihydroberberine, trans-resveratrol, ginger root extract, and methylcobalamin. Participants will take the provided supplement twice per day for the entire study duration in addition to pain management treatment protocols the participants currently follow.

SUMMARY:
This is a research study to evaluate the effectiveness of daily supplementation with Root.Health, a plant-based dietary supplement, on reducing levels of 11 abnormal urine biomarkers associated with chronic pain. Biomarkers are molecules found in blood, tissues, or other body fluids (such as urine) that indicate normal or abnormal processes.

DETAILED DESCRIPTION:
This study aims to utilize pain-specific abnormal biomarkers to evaluate how daily supplementation with Root.Health, a plant-based dietary supplement, affects FPI urine screening scores in chronic opioid-consuming pain patients. Analyzing the effect of Root.Health supplementation on pain-specific biomarkers through changes in FPI scores may expand our understanding of the degree to which these biomarkers may correlate to the underlying biologic processes involved in chronic pain creation. While widespread identification of such abnormalities may prove to have profound impacts on the future prevention, diagnosis, and treatment of pain, this investigation only intends to evaluate the effect of Root.Health on patient's urine levels of abnormal biomarkers. A previous validation study of the urine assay used in FPI screening demonstrated that an estimated 86% of patients reporting pain have at least one abnormal pain-related biomarker. The plant-based ingredients of the Root.Health supplement have been previously studied in the context of biochemical abnormalities that drive pain development, and this study is designed to characterize the mechanism by which these ingredients act to maintain biochemical processes which normally attenuate pain. As such, this study is not intended to evaluate Root.Health's ability to diagnose, cure, mitigate, treat, or prevent any disease.

The compounds included Root.Health supplements were carefully selected based on methodological review of current scientific evidence describing their roles in supporting innate physiological processes that attenuate biochemical abnormalities driving pain development. The investigators hypothesize that the plant-based compounds included in Root.Health will reduce the levels of abnormal pain biomarkers in chronic pain patients, as measured by a change in FPI score from baseline, based on literature which suggests that these compounds may attenuate biochemical abnormalities involved in causative pain mechanisms by supporting specific markers of cellular health (i.e normal activity of inflammatory pathways, oxidative stress capacity, production of pain-related neurotransmitters, and micronutrient status).

This is an open-label, prospective, observational pilot study. The investigators will be using a single group assignment intervention model with one group of 20 subjects. The primary outcome of this study is to evaluate Foundational Pain Index scores following a 3-month daily supplementation course with Root.Health in an opiate-using chronic pain patient population at 1-month and 3-months. The secondary objective of this study is to evaluate if daily supplementation with Root.Health for a 3-month study period affects Brief Pain Inventory (BPI) Short Form and Oswestry Disability Index (ODI) scores and/or opiate consumption in this patient population. The total study duration for each eligible participant is 4 months, which will include 5 study points: initial in-person study visit, 1-week in-person follow up visit (where study participants will receive supplements), and 3 virtual follow up visits at 1-month, 2-months and 3-months.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years of age or older
* At least two (2) or more symptoms of moderate or higher severity musculoskeletal pain for at least one year prior to study enrollment
* At least 3 months of opioid use for pain management at time of study enrollment

Exclusion Criteria:

* under 18 years of age
* participants who are pregnant or breastfeeding at time of study recruitment
* To reduce the likelihood of a study population whose recreational choices may affect the study endpoints, the investigators will screen potential participants during the enrollment phase using exclusion criteria based on health history, including recreational opiate drug use.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-08-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Effects on Foundation Pain Index (FPI) scores | 3 months
  To determine if a 3-month Root.Health supplementation course changes urine levels of Foundation Pain Index (FPI) scores mechanistic pain biomarkers in an opiate-using chronic pain population. Previous validation studies have demonstrated that higher FPI scores, represented by a greater number of abnormal biomarkers, indicate abnormal biochemical function is more likely to contribute to painful symptoms. Lower FPI scores, represented by a lower number of abnormal biomarkers, indicate biochemical function is unremarkable and is therefore less likely to be a contributor to painful symptoms. As such, the investigators will only include study participants with baseline FPI scores between 20-100 to select a study population in which abnormal biochemical functioning is more likely to be contributing to chronic pain symptoms. Scores between 0-20 are considered unremarkable.

SECONDARY OUTCOMES:
Pain Improvements | 3 months
  To evaluate if a 3-month Root.Health supplementation regimen changes Brief Pain Inventory (BPI) Short Form scores from time of study enrollment in an opiate-using chronic pain population. These tests are included in the standard of care for chronic pain patients.
  For each item of the BPI, patients select a whole number on scale of 0-10, where 0 indicates no pain and 10 indicates worst possible pain. Lower scores are associated with less severe episodes of pain.
Functional Improvements | 3 months
  To evaluate if a 3-month Root.Health supplementation regimen changes Oswestry Disability Index (ODI) scores from time of study enrollment in an opiate-using chronic pain population. These tests are included in the standard of care for chronic pain patients.
  For each question on the ODI, patient select the one whole number that describes how much the pain has interfered with the listed activities. The ODI is scored on a scale of 0-10, where 0 indicates no interference thus being able to do all activities and 10 indicates complete interference so the patient is unable to do the activity. Lower scores are associated with less severe episodes of pain.
Reduced Opioid Dependency | 3 months
  To evaluate if a 3-month Root.Health supplementation regimen affects opiate consumption habits from time of study enrollment in an opiate-using chronic pain population. This information will be gathered through subjective patient interviews at each month's follow up, inquiring about how often the patient is taking a prescribed medication. The study participants will report if they have continued their opioid medications at regular intervals as prescribed, or if they have taken less or more than the maximum prescribed dose.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathann Kuo, MD, Principal Investigator — Medical Director, Hudson Medical
Locations (1):
- Hudson Medical, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abbud W, Habinowski S, Zhang JZ, Kendrew J, Elkairi FS, Kemp BE, Witters LA, Ismail-Beigi F. Stimulation of AMP-activated protein kinase (AMPK) is associated with enhancement of Glut1-mediated glucose transport. Arch Biochem Biophys. 2000 Aug 15;380(2):347-52. doi: 10.1006/abbi.2000.1935. PMID 10933890
- [Background] Al Amin ASM, Gupta V. Vitamin B12 (Cobalamin). 2023 Jul 16. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK559132/ PMID 32644558
- [Background] Allen LH. Vitamin B-12. Adv Nutr. 2012 Jan;3(1):54-5. doi: 10.3945/an.111.001370. Epub 2012 Jan 5. No abstract available. PMID 22332101
- [Background] Aggarwal BB, Shishodia S. Molecular targets of dietary agents for prevention and therapy of cancer. Biochem Pharmacol. 2006 May 14;71(10):1397-421. doi: 10.1016/j.bcp.2006.02.009. Epub 2006 Feb 23. PMID 16563357
- [Background] Aggarwal BB, Harikumar KB. Potential therapeutic effects of curcumin, the anti-inflammatory agent, against neurodegenerative, cardiovascular, pulmonary, metabolic, autoimmune and neoplastic diseases. Int J Biochem Cell Biol. 2009 Jan;41(1):40-59. doi: 10.1016/j.biocel.2008.06.010. Epub 2008 Jul 9. PMID 18662800
- [Background] Amirdelfan K, Pope JE, Gunn J, Hill MM, Cotten BM, Beresh JE, Dobecki D, Miller N, Mehta P, Girardi G, Deer TR. Clinical Validation of a Multi-Biomarker Assay for the Evaluation of Chronic Pain Patients in a Cross-Sectional, Observational Study. Pain Ther. 2020 Dec;9(2):511-529. doi: 10.1007/s40122-020-00175-3. Epub 2020 Jun 3. PMID 32495188
- [Background] Anh NH, Kim SJ, Long NP, Min JE, Yoon YC, Lee EG, Kim M, Kim TJ, Yang YY, Son EY, Yoon SJ, Diem NC, Kim HM, Kwon SW. Ginger on Human Health: A Comprehensive Systematic Review of 109 Randomized Controlled Trials. Nutrients. 2020 Jan 6;12(1):157. doi: 10.3390/nu12010157. PMID 31935866
- [Background] Bailey RL, Jun S, Murphy L, Green R, Gahche JJ, Dwyer JT, Potischman N, McCabe GP, Miller JW. High folic acid or folate combined with low vitamin B-12 status: potential but inconsistent association with cognitive function in a nationally representative cross-sectional sample of US older adults participating in the NHANES. Am J Clin Nutr. 2020 Dec 10;112(6):1547-1557. doi: 10.1093/ajcn/nqaa239. PMID 32860400
- [Background] Asahi T, Wu X, Shimoda H, Hisaka S, Harada E, Kanno T, Nakamura Y, Kato Y, Osawa T. A mushroom-derived amino acid, ergothioneine, is a potential inhibitor of inflammation-related DNA halogenation. Biosci Biotechnol Biochem. 2016;80(2):313-7. doi: 10.1080/09168451.2015.1083396. Epub 2015 Sep 4. PMID 26338495
- [Background] Bannister K, Dickenson AH. What do monoamines do in pain modulation? Curr Opin Support Palliat Care. 2016 Jun;10(2):143-8. doi: 10.1097/SPC.0000000000000207. PMID 27043287
- [Background] Benson KF, Ager DM, Landes B, Aruoma OI, Jensen GS. Improvement of joint range of motion (ROM) and reduction of chronic pain after consumption of an ergothioneine-containing nutritional supplement. Prev Med. 2012 May;54 Suppl:S83-9. doi: 10.1016/j.ypmed.2012.02.001. Epub 2012 Feb 9. PMID 22342951
- [Background] Calvo MS, Mehrotra A, Beelman RB, Nadkarni G, Wang L, Cai W, Goh BC, Kalaras MD, Uribarri J. A Retrospective Study in Adults with Metabolic Syndrome: Diabetic Risk Factor Response to Daily Consumption of Agaricus bisporus (White Button Mushrooms). Plant Foods Hum Nutr. 2016 Sep;71(3):245-51. doi: 10.1007/s11130-016-0552-7. PMID 27193019
- [Background] Cheah IK, Halliwell B. Ergothioneine; antioxidant potential, physiological function and role in disease. Biochim Biophys Acta. 2012 May;1822(5):784-93. doi: 10.1016/j.bbadis.2011.09.017. Epub 2011 Oct 4. PMID 22001064
- [Background] Cheah IK, Tang RM, Yew TS, Lim KH, Halliwell B. Administration of Pure Ergothioneine to Healthy Human Subjects: Uptake, Metabolism, and Effects on Biomarkers of Oxidative Damage and Inflammation. Antioxid Redox Signal. 2017 Feb 10;26(5):193-206. doi: 10.1089/ars.2016.6778. Epub 2016 Sep 7. PMID 27488221
- [Background] Cheah IK, Halliwell B. Ergothioneine, recent developments. Redox Biol. 2021 Jun;42:101868. doi: 10.1016/j.redox.2021.101868. Epub 2021 Jan 26. PMID 33558182
- [Background] Chen JS, Alfajaro MM, Chow RD, Wei J, Filler RB, Eisenbarth SC, Wilen CB. Non-steroidal anti-inflammatory drugs dampen the cytokine and antibody response to SARS-CoV-2 infection. J Virol. 2021 Mar 10;95(7):e00014-21. doi: 10.1128/JVI.00014-21. Epub 2021 Jan 13. PMID 33441348
- [Background] Djade CD, Diorio C, Laurin D, Dionne CE. An exploratory identification of biological markers of chronic musculoskeletal pain in the low back, neck, and shoulders. PLoS One. 2022 Apr 15;17(4):e0266999. doi: 10.1371/journal.pone.0266999. eCollection 2022. PMID 35427389
- [Background] Stretanski MF, Kopitnik NL, Matha A, Conermann T. Chronic Pain. 2025 Sep 28. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK553030/ PMID 31971706
- [Background] Ehmedah A, Nedeljkovic P, Dacic S, Repac J, Draskovic Pavlovic B, Vucevic D, Pekovic S, Bozic Nedeljkovic B. Vitamin B Complex Treatment Attenuates Local Inflammation after Peripheral Nerve Injury. Molecules. 2019 Dec 17;24(24):4615. doi: 10.3390/molecules24244615. PMID 31861069
- [Background] Farah S, Yammine K. A systematic review on the efficacy of vitamin B supplementation on diabetic peripheral neuropathy. Nutr Rev. 2022 Apr 8;80(5):1340-1355. doi: 10.1093/nutrit/nuab116. PMID 34990506
- [Background] Feng R, Shou JW, Zhao ZX, He CY, Ma C, Huang M, Fu J, Tan XS, Li XY, Wen BY, Chen X, Yang XY, Ren G, Lin Y, Chen Y, You XF, Wang Y, Jiang JD. Transforming berberine into its intestine-absorbable form by the gut microbiota. Sci Rep. 2015 Jul 15;5:12155. doi: 10.1038/srep12155. PMID 26174047
- [Background] Gonzales AM, Orlando RA. Curcumin and resveratrol inhibit nuclear factor-kappaB-mediated cytokine expression in adipocytes. Nutr Metab (Lond). 2008 Jun 12;5:17. doi: 10.1186/1743-7075-5-17. PMID 18549505
- [Background] Gunn J, Hill MM, Cotten BM, Deer TR. An Analysis of Biomarkers in Patients with Chronic Pain. Pain Physician. 2020 Jan;23(1):E41-E49. PMID 32013287
- [Background] Gupta SC, Sung B, Kim JH, Prasad S, Li S, Aggarwal BB. Multitargeting by turmeric, the golden spice: From kitchen to clinic. Mol Nutr Food Res. 2013 Sep;57(9):1510-28. doi: 10.1002/mnfr.201100741. Epub 2012 Aug 13. PMID 22887802
- [Background] Habib SH, Makpol S, Abdul Hamid NA, Das S, Ngah WZ, Yusof YA. Ginger extract (Zingiber officinale) has anti-cancer and anti-inflammatory effects on ethionine-induced hepatoma rats. Clinics (Sao Paulo). 2008 Dec;63(6):807-13. doi: 10.1590/s1807-59322008000600017. PMID 19061005
- [Background] Hagedorn JM, Gunn J, Budwany R, D'Souza RS, Chakravarthy K, Deer TR. How Well Do Current Laboratory Biomarkers Inform Clinical Decision-Making in Chronic Pain Management? J Pain Res. 2021 Dec 3;14:3695-3710. doi: 10.2147/JPR.S311974. eCollection 2021. PMID 34887680
- [Background] Fu TT, Shen L. Ergothioneine as a Natural Antioxidant Against Oxidative Stress-Related Diseases. Front Pharmacol. 2022 Mar 18;13:850813. doi: 10.3389/fphar.2022.850813. eCollection 2022. PMID 35370675
- [Background] Halliwell B, Cheah IK, Tang RMY. Ergothioneine - a diet-derived antioxidant with therapeutic potential. FEBS Lett. 2018 Oct;592(20):3357-3366. doi: 10.1002/1873-3468.13123. Epub 2018 Jun 15. PMID 29851075
- [Background] Hosseinzadeh H, Moallem SA, Moshiri M, Sarnavazi MS, Etemad L. Anti-nociceptive and anti-inflammatory effects of cyanocobalamin (vitamin B12) against acute and chronic pain and inflammation in mice. Arzneimittelforschung. 2012 Jul;62(7):324-9. doi: 10.1055/s-0032-1311635. Epub 2012 May 15. PMID 22588629
- [Background] Jung YP, Earnest CP, Koozehchian M, Galvan E, Dalton R, Walker D, Rasmussen C, Murano PS, Greenwood M, Kreider RB. Effects of acute ingestion of a pre-workout dietary supplement with and without p-synephrine on resting energy expenditure, cognitive function and exercise performance. J Int Soc Sports Nutr. 2017 Jan 12;14:3. doi: 10.1186/s12970-016-0159-2. eCollection 2017. PMID 28096758
- [Background] Kumar S, Ahuja V, Sankar MJ, Kumar A, Moss AC. Curcumin for maintenance of remission in ulcerative colitis. Cochrane Database Syst Rev. 2012 Oct 17;10:CD008424. doi: 10.1002/14651858.CD008424.pub2. PMID 23076948
- [Background] Kunnumakkara AB, Bordoloi D, Padmavathi G, Monisha J, Roy NK, Prasad S, Aggarwal BB. Curcumin, the golden nutraceutical: multitargeting for multiple chronic diseases. Br J Pharmacol. 2017 Jun;174(11):1325-1348. doi: 10.1111/bph.13621. Epub 2016 Oct 21. PMID 27638428
- [Background] Lam-Sidun D, Peters KM, Borradaile NM. Mushroom-Derived Medicine? Preclinical Studies Suggest Potential Benefits of Ergothioneine for Cardiometabolic Health. Int J Mol Sci. 2021 Mar 23;22(6):3246. doi: 10.3390/ijms22063246. PMID 33806754
- [Background] Li L, Li J, Gao M, Fan H, Wang Y, Xu X, Chen C, Liu J, Kim J, Aliyari R, Zhang J, Jin Y, Li X, Ma F, Shi M, Cheng G, Yang H. Interleukin-8 as a Biomarker for Disease Prognosis of Coronavirus Disease-2019 Patients. Front Immunol. 2021 Jan 8;11:602395. doi: 10.3389/fimmu.2020.602395. eCollection 2020. PMID 33488599
- [Background] Li J, Zhang CX, Liu YM, Chen KL, Chen G. A comparative study of anti-aging properties and mechanism: resveratrol and caloric restriction. Oncotarget. 2017 Aug 9;8(39):65717-65729. doi: 10.18632/oncotarget.20084. eCollection 2017 Sep 12. PMID 29029466
- [Background] Liu T, Zhang L, Joo D, Sun SC. NF-kappaB signaling in inflammation. Signal Transduct Target Ther. 2017;2:17023-. doi: 10.1038/sigtrans.2017.23. Epub 2017 Jul 14. PMID 29158945
- [Background] Majeed M, Majeed S, Nagabhushanam K. Efficacy and Safety of Tetrahydrocurcuminoids for the Treatment of Canker Sore and Gingivitis. Evid Based Complement Alternat Med. 2020 Dec 16;2020:6611877. doi: 10.1155/2020/6611877. eCollection 2020. PMID 33381205
- [Background] Maroon JC, Bost JW, Maroon A. Natural anti-inflammatory agents for pain relief. Surg Neurol Int. 2010 Dec 13;1:80. doi: 10.4103/2152-7806.73804. PMID 21206541
- [Background] Mashhadi NS, Ghiasvand R, Askari G, Hariri M, Darvishi L, Mofid MR. Anti-oxidative and anti-inflammatory effects of ginger in health and physical activity: review of current evidence. Int J Prev Med. 2013 Apr;4(Suppl 1):S36-42. PMID 23717767
- [Background] Mobasheri A, Henrotin Y, Biesalski HK, Shakibaei M. Scientific evidence and rationale for the development of curcumin and resveratrol as nutraceutricals for joint health. Int J Mol Sci. 2012;13(4):4202-4232. doi: 10.3390/ijms13044202. Epub 2012 Mar 30. PMID 22605974
- [Background] Moon JM, Ratliff KM, Hagele AM, Stecker RA, Mumford PW, Kerksick CM. Absorption Kinetics of Berberine and Dihydroberberine and Their Impact on Glycemia: A Randomized, Controlled, Crossover Pilot Trial. Nutrients. 2021 Dec 28;14(1):124. doi: 10.3390/nu14010124. PMID 35010998
- [Background] Nakamura Y, Ohto Y, Murakami A, Osawa T, Ohigashi H. Inhibitory effects of curcumin and tetrahydrocurcuminoids on the tumor promoter-induced reactive oxygen species generation in leukocytes in vitro and in vivo. Jpn J Cancer Res. 1998 Apr;89(4):361-70. doi: 10.1111/j.1349-7006.1998.tb00572.x. PMID 9617340
- [Background] Park JS, Park D, Ko PW, Kang K, Lee HW. Serum methylmalonic acid correlates with neuropathic pain in idiopathic Parkinson's disease. Neurol Sci. 2017 Oct;38(10):1799-1804. doi: 10.1007/s10072-017-3056-9. Epub 2017 Jul 19. PMID 28726051
- [Background] Peabody JW, Luck J, Glassman P, Jain S, Hansen J, Spell M, Lee M. Measuring the quality of physician practice by using clinical vignettes: a prospective validation study. Ann Intern Med. 2004 Nov 16;141(10):771-80. doi: 10.7326/0003-4819-141-10-200411160-00008. PMID 15545677
- [Background] Pourhabibi-Zarandi F, Shojaei-Zarghani S, Rafraf M. Curcumin and rheumatoid arthritis: A systematic review of literature. Int J Clin Pract. 2021 Oct;75(10):e14280. doi: 10.1111/ijcp.14280. Epub 2021 May 24. PMID 33914984
- [Background] Qu H, Guo M, Chai H, Wang WT, Gao ZY, Shi DZ. Effects of Coenzyme Q10 on Statin-Induced Myopathy: An Updated Meta-Analysis of Randomized Controlled Trials. J Am Heart Assoc. 2018 Oct 2;7(19):e009835. doi: 10.1161/JAHA.118.009835. PMID 30371340
- [Background] Rahman I, Gilmour PS, Jimenez LA, Biswas SK, Antonicelli F, Aruoma OI. Ergothioneine inhibits oxidative stress- and TNF-alpha-induced NF-kappa B activation and interleukin-8 release in alveolar epithelial cells. Biochem Biophys Res Commun. 2003 Mar 21;302(4):860-4. doi: 10.1016/s0006-291x(03)00224-9. PMID 12646250
- [Background] Rosenblum A, Marsch LA, Joseph H, Portenoy RK. Opioids and the treatment of chronic pain: controversies, current status, and future directions. Exp Clin Psychopharmacol. 2008 Oct;16(5):405-16. doi: 10.1037/a0013628. PMID 18837637
- [Background] Sharifi-Rad J, Rayess YE, Rizk AA, Sadaka C, Zgheib R, Zam W, Sestito S, Rapposelli S, Neffe-Skocinska K, Zielinska D, Salehi B, Setzer WN, Dosoky NS, Taheri Y, El Beyrouthy M, Martorell M, Ostrander EA, Suleria HAR, Cho WC, Maroyi A, Martins N. Turmeric and Its Major Compound Curcumin on Health: Bioactive Effects and Safety Profiles for Food, Pharmaceutical, Biotechnological and Medicinal Applications. Front Pharmacol. 2020 Sep 15;11:01021. doi: 10.3389/fphar.2020.01021. eCollection 2020. PMID 33041781
- [Background] Shakibaei M, John T, Schulze-Tanzil G, Lehmann I, Mobasheri A. Suppression of NF-kappaB activation by curcumin leads to inhibition of expression of cyclo-oxygenase-2 and matrix metalloproteinase-9 in human articular chondrocytes: Implications for the treatment of osteoarthritis. Biochem Pharmacol. 2007 May 1;73(9):1434-45. doi: 10.1016/j.bcp.2007.01.005. Epub 2007 Jan 7. PMID 17291458
- [Background] Sforzini L, Nettis MA, Mondelli V, Pariante CM. Inflammation in cancer and depression: a starring role for the kynurenine pathway. Psychopharmacology (Berl). 2019 Oct;236(10):2997-3011. doi: 10.1007/s00213-019-05200-8. Epub 2019 Feb 26. PMID 30806743
- [Background] Staats Pires A, Heng B, Tan VX, Latini A, Russo MA, Santarelli DM, Bailey D, Wynne K, O'Brien JA, Guillemin GJ, Austin PJ. Kynurenine, Tetrahydrobiopterin, and Cytokine Inflammatory Biomarkers in Individuals Affected by Diabetic Neuropathic Pain. Front Neurosci. 2020 Aug 21;14:890. doi: 10.3389/fnins.2020.00890. eCollection 2020. PMID 32973438
- [Background] Tan L, Wang Y, Ai G, Luo C, Chen H, Li C, Zeng H, Xie J, Chen J, Su Z. Dihydroberberine, a hydrogenated derivative of berberine firstly identified in Phellodendri Chinese Cortex, exerts anti-inflammatory effect via dual modulation of NF-kappaB and MAPK signaling pathways. Int Immunopharmacol. 2019 Oct;75:105802. doi: 10.1016/j.intimp.2019.105802. Epub 2019 Aug 8. PMID 31401380
- [Background] Tian X, Cioccoloni G, Sier JH, Naseem KM, Thorne JL, Moore JB. Ergothioneine supplementation in people with metabolic syndrome (ErgMS): protocol for a randomised, double-blind, placebo-controlled pilot study. Pilot Feasibility Stud. 2021 Oct 29;7(1):193. doi: 10.1186/s40814-021-00929-6. PMID 34715934
- [Background] Wahab A, Gao K, Jia C, Zhang F, Tian G, Murtaza G, Chen J. Significance of Resveratrol in Clinical Management of Chronic Diseases. Molecules. 2017 Aug 18;22(8):1329. doi: 10.3390/molecules22081329. PMID 28820474
- [Background] Yin J, Xing H, Ye J. Efficacy of berberine in patients with type 2 diabetes mellitus. Metabolism. 2008 May;57(5):712-7. doi: 10.1016/j.metabol.2008.01.013. PMID 18442638
- [Background] Zhang JM, An J. Cytokines, inflammation, and pain. Int Anesthesiol Clin. 2007 Spring;45(2):27-37. doi: 10.1097/AIA.0b013e318034194e. PMID 17426506
- [Background] Zhang M, Han W, Hu S, Xu H. Methylcobalamin: a potential vitamin of pain killer. Neural Plast. 2013;2013:424651. doi: 10.1155/2013/424651. Epub 2013 Dec 26. PMID 24455309
- [Background] Zykova TA, Zhu F, Zhai X, Ma WY, Ermakova SP, Lee KW, Bode AM, Dong Z. Resveratrol directly targets COX-2 to inhibit carcinogenesis. Mol Carcinog. 2008 Oct;47(10):797-805. doi: 10.1002/mc.20437. PMID 18381589